CLINICAL TRIAL: NCT02102659
Title: This Preliminary Study Was Designed to Explore a New Biological Method for Nutritional Assessment by Measuring Oral Mucosal Epithelial Cell Apoptosis Rate and Guideline to Clinical Nutrition Support Therapy for Improving Clinical Outcome of Malnourished Patients.
Brief Title: Biological Assessment of Clinical Nutrition and Its Application
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jianping Gong, Director of Department of General Surgery, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJ-20130803
Record Dates: First submitted 2013-11-27; First posted 2014-04-03 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-03

CONDITIONS: Malnutrition
Keywords: Nutritional Assessment; Oral Epithelial Cell; Apoptosis
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Upper Limit Nutrition Support Therapy (Experimental): "Upper limit nutrition support therapy" will be used in patens assigned to this group based on the patient's curve of apoptosis of oral mucosal epithelium.
  Interventions: Genetic: Upper Limit Nutrition Support Therapy
- Formula Nutrition Support Therapy (Active Comparator): "Formula nutrition support therapy" will be used in patens assigned in this group based on Harris Bendiest Formula.
  Interventions: Genetic: Formula Nutrition Support Therapy

INTERVENTIONS:
Genetic: Upper Limit Nutrition Support Therapy — "Upper limit nutrition support therapy" will be used in patens assigned to this group based on the patient's curve of apoptosis of oral mucosal epithelium
  Other Names: Apoptosis rate of human oral epithelial cells
  Arms: Upper Limit Nutrition Support Therapy
Genetic: Formula Nutrition Support Therapy — "Formula nutrition support therapy" will be used in patens assigned in this group based on Harris Bendiest Formula.
  Arms: Formula Nutrition Support Therapy

SUMMARY:
1. Clinical nutritional support therapy is an important progress of modern medicine.
2. Conventional methods of clinical nutrition assessment (Anthropometric, lab, etc.) not just lack of accuracy and immediacy but also difficult to dynamically reflect the fluctuation trend of nutrition status.
3. It has been reported that malnutrition affects proliferation and apoptosis of human cells in vivo. This preliminary study was initiated by the hypothesis that changes in nutritional status may be reflected rapidly in fast proliferating cells.
4. In the previous studies the investigators already found that apoptosis rate of oral mucosal epithelium could reflect changes in nutritional status.There were an obvious decreasing in apoptosis and proliferation rate of oral mucosal epithelium in malnourished patients.
5. Based on the patient's curve of apoptosis rate of oral mucosal epithelium, the plateau being achieved by increase the nutrition amount continuously, Maintain this amount of nutrition given until the end of treatment. The investigators call this amount of nutrition the "upper limit nutrition support therapy".
6. The patients applying for"upper limit nutrition support therapy" and "Formula nutrition support therapy" separately, comparing of the two methods influences on postoperative wound healing, postoperative complication rate ,inflammatory response, side effects of chemotherapy, hospital stays and hospitalization expenses.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Gastric cancer or colorectal cancer which confirmed by Preoperative pathology will be included.
2. Patients who are diagnosed as malnutrition according history, physical examination and Nutrition Risk Screening 2002 will be included.
3. patients who have digestive tract fistula because of operation complication will be included.
4. patients who need fast track recovery after colorectal cancer operation will be included.

Exclusion Criteria:

1. Patients who are diagnosed as Late stage (stage IV) gastric cancer or colorectal cancer and can not accomplish radical resection will be excluded.
2. Postoperative gastric cancer or colorectal cancer patients who is Unable to tolerate the chemotherapy or unable to complete the whole chemotherapy course will be excluded.
3. patients with Severe endocrine system disease such as diabetic mellitus, hyperthyroidism will be excluded.
4. patients with cardiac, renal, respiratory, or hepatic diseases, diabetes,active infection, evidence of sepsis, active bleeding or obstruction, and oral disease will be excluded.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 167 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
The Length and Width of Surgical Incision Edema | 2nd day
  The length and width of surgical incision edema will be measured by doppler ultrasonography in the 2nd day respectively after gastrointestinal operation.
The Length and Width of Surgical Incision Edema | 9th day
  The length and width of surgical incision edema will be measured by doppler ultrasonography in the 9th day respectively after gastrointestinal operation.

SECONDARY OUTCOMES:
Oral Mucosal Epithelial Cell Apoptosis Rate | 10 or 12 days
  Oral mucosal epithelial cell samples will be collected in the every morning before tooth brushing teeth for 9 days after gastrointestinal operation..The cells well be analyzed by flow cytometry for detecting apoptosis rate.
Anthropometric measurements | 9 days
  Anthropometric measurements including weight, body mass index, triceps skinfold thickness, and midarm muscle circumference will be recorded every 2-3 days days for 9 days after gastrointestinal operation..
The level of serum proteins | 9 days
  The serum proteins including retinol-binding protein (RBP), transferrin, prealbumin (PA), and albumin will be measured every 2-3 days for 9 days after gastrointestinal operation.

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Gong, M.D.,Ph.D., Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Tongji Medical College in Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Background] Studley HO. Percentage of weight loss: a basic indicator of surgical risk in patients with chronic peptic ulcer. 1936. Nutr Hosp. 2001 Jul-Aug;16(4):141-3; discussion 140-1. No abstract available. PMID 11680474
- [Background] Schiesser M, Muller S, Kirchhoff P, Breitenstein S, Schafer M, Clavien PA. Assessment of a novel screening score for nutritional risk in predicting complications in gastro-intestinal surgery. Clin Nutr. 2008 Aug;27(4):565-70. doi: 10.1016/j.clnu.2008.01.010. Epub 2008 Mar 17. PMID 18342995
- [Background] Norman K, Pichard C, Lochs H, Pirlich M. Prognostic impact of disease-related malnutrition. Clin Nutr. 2008 Feb;27(1):5-15. doi: 10.1016/j.clnu.2007.10.007. Epub 2007 Dec 3. PMID 18061312
- [Background] Jones JS, Tidwell B, Travis J, Spencer T, Phillips P, Burford B. Nutritional support of the hospitalized patient: a team approach. J Miss State Med Assoc. 1995 Apr;36(4):91-9. PMID 7776363
- [Background] Li C, Thompson CB. Cancer. DNA damage, deamidation, and death. Science. 2002 Nov 15;298(5597):1346-7. doi: 10.1126/science.1079168. No abstract available. PMID 12434041
- [Background] Gong J, Traganos F, Darzynkiewicz Z. A selective procedure for DNA extraction from apoptotic cells applicable for gel electrophoresis and flow cytometry. Anal Biochem. 1994 May 1;218(2):314-9. doi: 10.1006/abio.1994.1184. PMID 8074286
- [Result] Gao C, Hasan O, Wei X, Zou Y, Yin X, Tao D, Gong J. Assessment of nutritional status of clinical patients by determining normal range of oral mucosal apoptosis and proliferation rate. J Huazhong Univ Sci Technolog Med Sci. 2012 Oct;32(5):680-685. doi: 10.1007/s11596-012-1017-3. Epub 2012 Oct 18. PMID 23073796
- [Result] Luo X, Zhou Y, Tao D, Yu Y, Hu J, Qiu F, Kulkarni H, Gong J. Usefulness of oral mucosal epithelial cell apoptosis rate in nutritional assessment. Nutrition. 2006 Oct;22(10):1032-8. doi: 10.1016/j.nut.2006.03.016. Epub 2006 Sep 15. PMID 16979323